CLINICAL TRIAL: NCT04352543
Title: Metabolic, Cardiovascular and Psychological Responses to Active Video Game in Older Adults
Brief Title: Active Video Game on Metabolic, Cardiovascular, and Psychological Metrics in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giselle Soares Passos, Clinical Professor, Universidade Federal de Goias
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.750.982
Record Dates: First submitted 2020-03-18; First posted 2020-04-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Aging
Keywords: physical activity; active video game; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults group (Experimental): Group of older adults >60 years old.
  Interventions: Behavioral: Active Video Game Exercise; Behavioral: Treadmill walking exercise; Behavioral: Sedentary Behavior

INTERVENTIONS:
Behavioral: Active Video Game Exercise — Play during 30 minutes in the easy level
Behavioral: Treadmill walking exercise — 30 minutes (65 - 75% heart rate maximal)
Behavioral: Sedentary Behavior — Quiet Rest: 30 minutes

SUMMARY:
The Xbox Kinect seems to be a good alternative for the older adults to perform physical activities at times that are typically associated with sedentary behaviors. The Xbox Kinect active video game has been used in various parts of the world as entertainment. The study of metabolic, cardiovascular and psychological responses during these activities may bring relevant information regarding the intensity of the exercises and, consequently, about the possibility of using these games to maintain and / or improve the cardiorespiratory fitness of the older adults. In addition, the present study may clarify the responses of activities on Xbox Kinect in elderly people with anxiety and depression symptoms. Will be selected 100 older adults. All volunteers will initially perform assessments of resting metabolic rate, cardiorespiratory fitness, functional tests, as well as subjective assessments of physical activity level, anxiety and mood. Subsequently, they will perform activities with body movements on the Xbox Kinect, which will be compared with sedentary behavior activity (TV / Movie). All activities will be monitored by means of a gas analyzer, which will record information about the behavior of energy expenditure, resting heart rate and activity. In addition, assessments of perception of effort and fun during activities will be made through subjective scales. The effects of Xbox Kinect activity on anxiety symptoms and mood will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age > 60 years
* Mini-mental score ≥ 24
* non-smoker
* no beta-blockers
* no cardiovascular risk

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — >60 years old
Enrollment: 32 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Anxiety State at 5 min before, and 5 and 20 minutes following exercise | 5 min before, and 5 and 20 minutes following exercise
  Anxiety Inventory-STAI trait-state. The scale encompass 20 items and provides a one-dimensional measurement. The score varies from 20 to 80 points, with scores indicating low (0-30), medium (31-49) or high (50 or more) level of anxiety.
  of anxiety.
Change from Baseline Mood States at 5 min before, and 5 and 20 minutes following exercise | 5 min before, and 5 and 20 minutes following exercise
  Scale: Profile of mood states (POMS) The POMS questionnaire is an instrument to evaluate mood states. It has 65 items and 6 domains: tension-anxiety, depression, anger-hostility, vigour-activity, fatigue, and confusion- bewilderment. The total mood disturbance score is derived by subtracting the vigour-activity score from the the sum of scores from the other subscales
Change from Baseline Exercise Experience at 5 min before, and 5 and 20 minutes following exercise | 5 min before, and 5 and 20 minutes following exercise
  Subjective Exercise Experiences Scale - SEES is a set of three subscales objectives that add up to 12 adjectives in total. A subscale well-being positive is composed of the following adjectives: great, positive, vigorous and wonderful; an anguish of the subscale psychological is composed by the adjectives lousy, diminished, discouraged and sad; while in the fatigue subscale, adjectives are: exhausted, exhausted, fatigued and tired. Each adjective can be classified into certain intensities create scores that can range from 1 (which means "nothing") to 7 points (which means "a lot"). Of that Thus, a score on each subscale can be at least 4 and a maximum of 28 points.

SECONDARY OUTCOMES:
Assess of Dementia | baseline
  Mini-Mental Scale - The MMSE is divided into five subscales (orientation, immediate memory, attention and calculation, evocation and language) and is used to screen for clinical symptoms of dementia. The MMSE score can vary from a minimum of 0 to a maximum total of 30 points. The cut-off point for the exam is 24 points.
Evaluation of habitual physical activity | baseline
  International Physical Activity Questionnaire (IPAQ) -
  1. VERY ACTIVE: one who has fulfilled recommendations from:
     1. VIGOROUS: 5 days / week and 30 minutes for session and / or
     2. VIGOROUS: 3 days / week and 20 minutes per + MODERATE and / or WALK session: 5 days / week and 30 minutes per session.
  2. ACTIVE: one who has followed the recommendations in:
     1. VIGOROUS: 3 days / week and 20 minutes per session; and / or
     2. MODERATE or WALK: 5 days / week and 30 minutes per session; and / or
     3. Any combined activity: 5 days / week and 150 minutes / week (walking + moderate + vigorous).
  3. IRREGULATELY ACTIVE: one who performs physical activity, but insufficient to be classified as active, as it does not comply with the recommendations frequency or duration.
  4. SEDENTARY: one who did not perform no physical activity for at least 10 minutes during the week.
Evaluation of Quality of Life | baseline
  SF-36 Short-Form - The SF-36 is a multidimensional questionnaire that covers eight components: physical functioning, role limitations due to physical health problems, role limitations due to emotional health problems, social functioning, vitality, general health perception, body pain, and mental health. All scores ranged from 0 to 100, with a higher score indicating better quality of life.
Evaluation of depression | baseline
  15-item Geriatric Depression Scale (GDS-15) is used to assess depressive symptoms. Participants who scored a total of 7 or more points are defined as having clinically significant depressive symptoms. The severity of depressive symptoms are: no depression (score of 0), questionable depression (score of 1-4), mild-to-moderate depression (score of 5-9) and severe depression (score of 10-15).
Evaluation of Anxiety trait | baseline
  Trait Anxiety (STAI) - The scale encompass 20 items and provides a one-dimensional measurement. The score varies from 20 to 80 points, with scores indicating low (0-30), medium (31-49) or high (50 or more) level of anxiety.
Medical Screening | baseline
  Clinical evaluation - patient's health history is registered. Previous disorders.
Cardiopulmonary exercise testing | baseline
  Bruce Protocol by FitMateTM Pro (Cosmed, Italy) will be used to obtain VO2max
Stress electrocardiogram (ECG) | baseline
  Bruce Protocol will be used. The exam will report the presence or absence of cardiovascular disease (exclusion criteria of the study)
Anthropometric Evaluation | baseline
  BMI
Evaluation of Resting Metabolic Rate | baseline
  Energy cost by FitMateTM Pro (Cosmed, Italy)
Anxiety symptoms | baseline
  Geriatric Anxiety Inventory: The GAI is a 20-item measure of anxiety symptoms severity developed for older adults. Scores ≥ 8 indicate the presence of anxiety symptoms.
6-Min Walk Test | baseline
  The 6-MWT is performed in a 20-m-long indoor hallway free of obstacles. Participants are instructed to walk at a self-selected regular pace to cover as much distance as they could during the allotted time. The score is the total number of meters walked in 6 min
8-ft Timed Up & Go Test (TUG) | baseline
  The 8-ft Timed Up & Go Test is used to assess agility and dynamic balance. Participants are asked to sito n a chair. On cue, they stood up, walked as quickly as possible around a cone set 8ft from the chair, and sat back down on the chair. Total time to complete the test in seconds was measured to assess performance.
Chair-Stand Test (CS) | baseline
  Chair Stand Test is used to assess lower body strength. After a signal participants completed as many "stand-ups" as possible with 30s. Total repetitions completed within 30s are used to score the participants' performance.
Chair sit-and-reach Test | baseline
  Chair sit-and-reach is used to evaluate lower body flexibility. Participants are asked to sit on the edge of a chair with the knee bent at 900 and the left foot flat on the while keeping the right knee straight and right leg extended forward. Participants are asked to attempt to touch their toes using both hands. The distance in inches between fingers and toes was measured and given a negative value if the fingers did not reach the toes and a positive value if fingers extended beyond the toes.
Metabolic assessment - Energy cost (joules/min) | baseline
  * Sedentary behavior (Watching Film/TV): 10 min
  * Active behavior (Playing Xbox Kinect): 10 min activity by 5 min rest (5 activities)FitMateTM Pro (Cosmed, Italy).
Heart rate (bpm) | baseline
  * Sedentary behavior (Watching Film/TV): 10 min
  * Active behavior (Playing Xbox Kinect): 10 min activity by 5 min rest (5 activities)FitMateTM Pro (Cosmed, Italy).
VO2 (ml/kg/min) | baseline
  * Sedentary behavior (Watching Film/TV): 10 min
  * Active behavior (Playing Xbox Kinect): 10 min activity by 5 min rest (5 activities)FitMateTM Pro (Cosmed, Italy).
Evaluation of Enjoyment | baseline
  PACES - consisting of five items. Each item has a score from 1 to 7 on a Likert scale. The sum of these items generates a range of scores from 5 to 35. Higher scores indicate greater enjoyment. The scores were transformed into percentage, with a score of 35 equal to 100%.
  * Sedentary behavior (Watching Film/TV): 10 min
  * Active behavior (Playing Xbox Kinect): 10 min activity by 5 min rest (5 activities)
Subjective perceived exertion | baseline
  The Borg Scale is used to verify the subjective perception of effort. This scale has 15 points, from 6 to 20. Each number refers to a certain intensity, so that the exercise can be classified as: no effort (6), extremely light (7), very light (8 and 9) , light (10 and 11), moderate (12 and 13), intense (14 and 15), very intense (16 and 17), extremely intense (18 and 19) and maximum effort.
  * Sedentary behavior (Watching Film/TV): 10 min
  * Active behavior (Playing Xbox Kinect): 10 min activity by 5 min rest (5 activities)

CONTACTS AND LOCATIONS:
Locations (1):
- UFG, Jatai, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferreira JA, Passos GS, Youngstedt SD, de Lima BE, Vieira LB, Martins MM, de Assis BP, Santana MG. Are there sex differences in energy expenditure and enjoyment in older adults playing active video games? J Bodyw Mov Ther. 2022 Jul;31:72-76. doi: 10.1016/j.jbmt.2022.04.008. Epub 2022 Apr 19. PMID 35710225